CLINICAL TRIAL: NCT00343564
Title: A Phase I-II Study to Determine the Safety, Pharmacokinetics and Potential Efficacy of Intravenous Administration of SB-743921 on Days 1 and 15 of a 28-Day Dosing Schedule in Patients With Non-Hodgkin Lymphoma and Hodgkin Lymphoma
Brief Title: A Study of SB-743921 in Non-Hodgkin Lymphoma and Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CY 2121
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Results first posted 2016-10-04 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkin's Disease
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — SB 743921

ARMS (2):
- Phase 1 Dose Escalation (Experimental): Phase 1 dose escalation without and with GCSF support
  Interventions: Drug: SB-743921
- Phase 2 Fixed Dose (Experimental): Phase 2 fixed dose based on Phase I findings stratified by NHL type
  Interventions: Drug: SB-743921

INTERVENTIONS:
Drug: SB-743921 — Phase 1: I.V. dose on Days 1 and 15 of a 28 day cycle starting at 2mg/m2 and increasing by 1 mg/m2 with possible prophylactic granulopoietic support until unacceptable toxicity develops.
  Arms: Phase 1 Dose Escalation
Drug: SB-743921 — Phase 2: I.V. dose and regimen will be determined based on Phase 1 findings.
  Arms: Phase 2 Fixed Dose

SUMMARY:
This study was an early-phase trial arranged into two phases. The Phase I portion was a dose-escalation study designed to assess the safety, tolerability and to identify the maximum tolerated dose of SB-743921 in patients with Non-Hodgkin Lymphoma and Hodgkin Lymphoma. Phase II was intended to assess the activity, safety and tolerability of SB-743921 in patients with Indolent and Aggressive Non-Hodgkin's Lymphomas exclusively. The Phase II portion of the study was not initiated.

ELIGIBILITY:
Inclusion Criteria: Phase 1: Patients with evaluable or measurable (by MRI or CT) Hodgkin's Disease or Non-Hodgkin's Lymphoma. Phase 2: Patients with Measurable Non-Hodgkin's Lymphomas (Indolent or Aggressive) only. - Patients with Indolent NHL must be relapsed or refractory to at least one prior line of therapy (CHOP, CVP, chlorambucil or fludaribine). Prior treatment with Rituximab is required. - Patients with Aggressive NHL refractory to (or relapsed from) at least one CHOP-based therapy who have had prior treatment with Rituximab and who are not candidates for high-dose chemotherapy or autologous stem cell transplantation. - ECOG performance status 0-2 - Autologous stem cell transplant recipients are eligible if 100 days have elapsed since procedure. Exclusion Criteria: Phase 1: History of prior radioimmunotherapy (Bexxar, Zevalin); These patients ARE permitted in the Phase 2 trial. - Current active malignancy besides NHL, except excised non-melanoma skin cancer, in-situ cervical or bladder cancer or early stage prostate cancer. - Patients with leptomeningeal of CNS lymphoma - Known allergy to and/or receipt of treatments contraindicated by administration of G-CSF - Patients with active Hepatitis B or C, or patients with HIV infection. - Pregnant or breast-feeding females. - Previous treatment with a KSP inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2006-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Owen O'Connor, M.D./Ph.D., Principal Investigator — Columbia University
Locations (8):
- United States (6):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cornell University Medical Center, New York, New York
  - Memorial Sloan-Kettering Caner Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Sarah Cannon Cancer Research Institute, Nashville, Tennessee
- Russia (2):
  - Russian Medical Academy of Postgraduate Education, Moscow
  - St. Petersburg State PAVLOV Medical University, Saint Petersburg

REFERENCES:
- [Derived] O'Connor OA, Gerecitano J, Van Deventer H, Hainsworth J, Zullo KM, Saikali K, Seroogy J, Wolff A, Escandon R. The addition of granulocyte-colony stimulating factor shifts the dose limiting toxicity and markedly increases the maximum tolerated dose and activity of the kinesin spindle protein inhibitor SB-743921 in patients with relapsed or refractory lymphoma: results of an international, multicenter phase I/II study. Leuk Lymphoma. 2015;56(9):2585-91. doi: 10.3109/10428194.2015.1004167. Epub 2015 Sep 11. PMID 25665464

RESULTS

PARTICIPANT FLOW:
Groups:
- 2 mg/m2 Without GCSF: Phase 1 dose escalation cohort 1 without GCSF support
- 3 mg/m2 Without GCSF: Phase 1 dose escalation cohort 2 without GCSF support
- 4 mg/m2 Without GCSF: Phase 1 dose escalation cohort 3 without GCSF support
- 5 mg/m2 Without GCSF: Phase 1 dose escalation cohort 4 without GCSF support
- 6 mg/m2 Without GCSF: Phase 1 dose escalation cohort 5 without GCSF support
- 7 mg/m2 Without GCSF: Phase 1 dose escalation cohort 6 without GCSF support
- 6 mg/m2 With GCSF: Phase 1 dose escalation cohort 1 with GCSF support
- 7 mg/m2 With GCSF: Phase 1 dose escalation cohort 2 with GCSF support
- 8 mg/m2 With GCSF: Phase 1 dose escalation cohort 3 with GCSF support
- 9 mg/m2 With GCSF: Phase 1 dose escalation cohort 4 with GCSF support
- 10 mg/m2 With GCSF: Phase 1 dose escalation cohort 5 with GCSF support
Period: Overall Study
Arm/Group | 2 mg/m2 Without GCSF | 3 mg/m2 Without GCSF | 4 mg/m2 Without GCSF | 5 mg/m2 Without GCSF | 6 mg/m2 Without GCSF | 7 mg/m2 Without GCSF | 6 mg/m2 With GCSF | 7 mg/m2 With GCSF | 8 mg/m2 With GCSF | 9 mg/m2 With GCSF | 10 mg/m2 With GCSF
Started | 6 | 7 | 3 | 7 | 10 | 9 | 4 | 3 | 3 | 8 | 8
Completed | 6 | 7 | 3 | 7 | 10 | 9 | 4 | 3 | 3 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 mg/m2 Without GCSF | 3 mg/m2 Without GCSF | 4 mg/m2 Without GCSF | 5 mg/m2 Without GCSF | 6 mg/m2 Without GCSF | 7 mg/m2 Without GCSF | 6 mg/m2 With GCSF | 7 mg/m2 With GCSF | 8 mg/m2 With GCSF | 9 mg/m2 With GCSF | 10 mg/m2 With GCSF | Total
Number analyzed (Participants) | 6 | 7 | 3 | 7 | 10 | 9 | 4 | 3 | 3 | 8 | 8 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 4 | 7 | 3 | 3 | 8 | 6 | 1 | 2 | 1 | 4 | 4 | 43
  >=65 years | 2 | 0 | 0 | 4 | 2 | 2 | 3 | 1 | 2 | 4 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (9) | 43 (13) | 33 (9) | 57 (22) | 48 (16) | 42 (24) | 69 (12) | 63 (11) | 63 (17) | 48 (22) | 56 (20) | 52 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 1 | 2 | 4 | 4 | 2 | 1 | 1 | 3 | 1 | 29
  Male | 2 | 1 | 2 | 5 | 6 | 5 | 2 | 2 | 2 | 5 | 7 | 39
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 1 | 5 | 7 | 6 | 4 | 3 | 2 | 8 | 7 | 53
  Russian Federation | 0 | 3 | 2 | 2 | 3 | 3 | 0 | 0 | 1 | 0 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Determination of Maximum Tolerated Dose (MTD) First Without and Then With Administration of Prophylactic G-CSF.
Description: Maximum Tolerated Dose (MTD) was determined by testing increasing doses in cohorts with at least 3 patients each. MTD reflects the highest dose of drug that did not cause dose limiting toxicity (DLT).
Time Frame: 28 days
Population: Safety population; all patients who received at least 1 dose of study drug were included in the intent-to-treat/safety populations. Efficacy evaluable; any patient who received both cycles of treatment.
Measure: Number; unit: mg/m2
Groups:
- Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF); Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF); Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF); Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF); Dose Escalation Cohort 5 6 mg/m2 (w/o GCSF); Dose Escalation Cohort 6 7 mg/m2 (w/o GCSF): Maximum Tolerated Dose (MTD) was determined by testing increasing doses without GCSF support
- Dose Escalation Cohort 1 6 mg/m2 (w/ GCSF); Dose Escalation Cohort 2 7mg/m2 (w/GCSF); Dose Escalation Cohort 3 8 mg/m2 (w/GCSF); Dose Escalation Cohort 4 9 mg/m2 (w/GCSF); Dose Escalation Cohort 5 10 mg/m2 (w/GCSF): Maximum Tolerated Dose (MTD) was determined by testing increasing doses with GCSF support
Arm/Group | Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF) | Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF) | Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF) | Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF) | Dose Escalation Cohort 5 6 mg/m2 (w/o GCSF) | Dose Escalation Cohort 6 7 mg/m2 (w/o GCSF) | Dose Escalation Cohort 1 6 mg/m2 (w/ GCSF) | Dose Escalation Cohort 2 7mg/m2 (w/GCSF) | Dose Escalation Cohort 3 8 mg/m2 (w/GCSF) | Dose Escalation Cohort 4 9 mg/m2 (w/GCSF) | Dose Escalation Cohort 5 10 mg/m2 (w/GCSF)
Number analyzed (Participants) | 4 | 6 | 3 | 5 | 6 | 9 | 4 | 3 | 3 | 7 | 6
mg/m2 | 2 | 3 | 4 | 5 | 6 | 6 | 6 | 7 | 8 | 9 | 9

2. Secondary Outcome: Characterization of PK (Cmax) of SB-743921 Administered as a 1-hour Intravenous Infusion on Day 1
Time Frame: Pre-dose, immediately post-dose, between 2 and 4 hours post-dose and between 24 and 36 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF); Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF); Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF); Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF); Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 3 8 mg/m2 (w/GCSF); Dose Escalation Cohort 4 9 mg/m2 (w/GCSF); Dose Escalation Cohort 5 10 mg/m2 (w/GCSF): Day 1 Cmax
Arm/Group | Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF) | Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF) | Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF) | Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF) | Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 3 8 mg/m2 (w/GCSF) | Dose Escalation Cohort 4 9 mg/m2 (w/GCSF) | Dose Escalation Cohort 5 10 mg/m2 (w/GCSF)
Number analyzed (Participants) | 5 | 6 | 3 | 6 | 13 | 12 | 3 | 7 | 6
ng/mL | 172 (40.7) | 348 (86.6) | 357 (50.4) | 514 (177) | 600 (175) | 689 (401) | 1130 (189) | 805 (501) | 1180 (682)

3. Secondary Outcome: Characterization of PK (Tmax) of SB-743921 Administered as a 1-hour Intravenous Infusion on Day1
Time Frame: Pre-dose, immediately post-dose, between 2 and 4 hours post-dose and between 24 and 36 hours post-dose
Measure: Mean (Standard Deviation); unit: hr
Groups:
- Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF); Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF); Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF); Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF); Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 3 8 mg/m2 (w/GCSF); Dose Escalation Cohort 4 9 mg/m2 (w/GCSF); Dose Escalation Cohort 5 10 mg/m2 (w/GCSF): Day 1 Tmax
Arm/Group | Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF) | Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF) | Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF) | Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF) | Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 3 8 mg/m2 (w/GCSF) | Dose Escalation Cohort 4 9 mg/m2 (w/GCSF) | Dose Escalation Cohort 5 10 mg/m2 (w/GCSF)
Number analyzed (Participants) | 5 | 6 | 3 | 6 | 13 | 12 | 3 | 7 | 6
hr | 1.20 (0.45) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00) | 1.08 (0.28) | 1.00 (0.43) | 1.00 (0.00) | 1.00 (0.00) | 1.17 (0.41)

4. Secondary Outcome: Characterization of PK (Clast) of SB-743921 Administered as a 1-hour Intravenous Infusion on Day 1
Time Frame: Pre-dose, immediately post-dose, between 2 and 4 hours post-dose and between 24 and 36 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF); Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF); Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF); Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF); Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 3 8 mg/m2 (w/GCSF); Dose Escalation Cohort 4 9 mg/m2 (w/GCSF); Dose Escalation Cohort 5 10 mg/m2 (w/GCSF): Day 1 Clast
Arm/Group | Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF) | Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF) | Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF) | Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF) | Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 3 8 mg/m2 (w/GCSF) | Dose Escalation Cohort 4 9 mg/m2 (w/GCSF) | Dose Escalation Cohort 5 10 mg/m2 (w/GCSF)
Number analyzed (Participants) | 5 | 6 | 3 | 6 | 13 | 12 | 3 | 7 | 6
ng/mL | 36.9 (23.6) | 61.6 (29.4) | 59.5 (39.9) | 79.1 (51.9) | 133 (64.7) | 103 (48.3) | 144 (97.6) | 122 (69.6) | 245 (134)

5. Secondary Outcome: Characterization of PK (AUClast) of SB-743921 Administered as a 1-hour Intravenous Infusion on Day 1
Time Frame: Pre-dose, immediately post-dose, between 2 and 4 hours post-dose and between 24 and 36 hours post-dose
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF); Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF); Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF); Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF); Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 3 8 mg/m2 (w/GCSF); Dose Escalation Cohort 4 9 mg/m2 (w/GCSF); Dose Escalation Cohort 5 10 mg/m2 (w/GCSF): Day 1 AUClast
Arm/Group | Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF) | Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF) | Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF) | Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF) | Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 3 8 mg/m2 (w/GCSF) | Dose Escalation Cohort 4 9 mg/m2 (w/GCSF) | Dose Escalation Cohort 5 10 mg/m2 (w/GCSF)
Number analyzed (Participants) | 5 | 6 | 3 | 6 | 13 | 12 | 3 | 7 | 6
hr*ng/mL | 1807 (1104) | 2800 (988.6) | 3269 (950.2) | 3707 (1750) | 5838 (2588) | 5359 (3028) | 6270 (2751) | 5875 (3483) | 11570 (6318)

6. Secondary Outcome: Characterization of PK (Cmax) of SB-743921 Administered as a 1-hour Intravenous Infusion on Day 15
Time Frame: Pre-dose, immediately post-dose, between 2 and 4 hours post-dose and between 24 and 36 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF); Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF); Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF); Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF); Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 3 8 mg/m2 (w/GCSF); Dose Escalation Cohort 4 9 mg/m2 (w/GCSF); Dose Escalation Cohort 5 10 mg/m2 (w/GCSF): Day 15 Cmax
Arm/Group | Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF) | Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF) | Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF) | Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF) | Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 3 8 mg/m2 (w/GCSF) | Dose Escalation Cohort 4 9 mg/m2 (w/GCSF) | Dose Escalation Cohort 5 10 mg/m2 (w/GCSF)
Number analyzed (Participants) | 3 | 5 | 3 | 8 | 13 | 8 | 3 | 7 | 6
ng/mL | 220 (51.2) | 323 (120) | 365 (45.2) | 599 (383) | 717 (278) | 835 (442) | 685 (163) | 706 (344) | 1430 (1620)

7. Secondary Outcome: Characterization of PK (Tmax) of SB-743921 Administered as a 1-hour Intravenous Infusion on Day 15
Time Frame: Pre-dose, immediately post-dose, between 2 and 4 hours post-dose and between 24 and 36 hours post-dose
Measure: Mean (Standard Deviation); unit: hr
Groups:
- Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF); Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF); Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF); Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF); Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 3 8 mg/m2 (w/GCSF); Dose Escalation Cohort 4 9 mg/m2 (w/GCSF); Dose Escalation Cohort 5 10 mg/m2 (w/GCSF): Day 15 Tmax
Arm/Group | Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF) | Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF) | Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF) | Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF) | Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 3 8 mg/m2 (w/GCSF) | Dose Escalation Cohort 4 9 mg/m2 (w/GCSF) | Dose Escalation Cohort 5 10 mg/m2 (w/GCSF)
Number analyzed (Participants) | 3 | 5 | 3 | 8 | 13 | 8 | 3 | 7 | 6
hr | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00)

8. Secondary Outcome: Characterization of PK (Clast) of SB-743921 Administered as a 1-hour Intravenous Infusion on Day 15
Time Frame: Pre-dose, immediately post-dose, between 2 and 4 hours post-dose and between 24 and 36 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF); Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF); Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF); Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF); Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 3 8 mg/m2 (w/GCSF); Dose Escalation Cohort 4 9 mg/m2 (w/GCSF); Dose Escalation Cohort 5 10 mg/m2 (w/GCSF): Day 15 Clast
Arm/Group | Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF) | Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF) | Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF) | Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF) | Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 3 8 mg/m2 (w/GCSF) | Dose Escalation Cohort 4 9 mg/m2 (w/GCSF) | Dose Escalation Cohort 5 10 mg/m2 (w/GCSF)
Number analyzed (Participants) | 3 | 5 | 3 | 8 | 13 | 8 | 3 | 7 | 6
ng/mL | 29.2 (11.8) | 84.2 (60.8) | 58.5 (29.8) | 84.6 (47.9) | 138 (103) | 92.4 (50.5) | 138 (94.9) | 150 (105) | 285 (290)

9. Secondary Outcome: Characterization of PK (AUClast) of SB-743921 Administered as a 1-hour Intravenous Infusion on Day 15
Time Frame: Pre-dose, immediately post-dose, between 2 and 4 hours post-dose and between 24 and 36 hours post-dose
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF); Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF); Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF); Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF); Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF); Dose Escalation Cohort 3 8 mg/m2 (w/GCSF); Dose Escalation Cohort 4 9 mg/m2 (w/GCSF): Day 15 AUClast
Arm/Group | Dose Escalation Cohort 1 2 mg/m2 (w/o GCSF) | Dose Escalation Cohort 2 3 mg/m2 (w/o GCSF) | Dose Escalation Cohort 3 4 mg/m2 (w/o GCSF) | Dose Escalation Cohort 4 5 mg/m2 (w/o GCSF) | Dose Escalation Cohort 5 6 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 6 7 mg/m2 (w/ and w/o GCSF) | Dose Escalation Cohort 3 8 mg/m2 (w/GCSF) | Dose Escalation Cohort 4 9 mg/m2 (w/GCSF) | Dose Escalation Cohort 5 10 mg/m2 (w/GCSF)
Number analyzed (Participants) | 3 | 5 | 3 | 8 | 13 | 8 | 3 | 7 | 6
hr*ng/mL | 1809 (464.1) | 2363 (1187) | 3380 (1456) | 4105 (2190) | 5869 (3417) | 5116 (1728) | 6041 (3010) | 6178 (3630) | 12590 (17850)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 28-day treatment period and at a 14-day follow up visit.
Description: Patients who received at least 1 dose of treatment were considered eligible for safety.
Arm/Group | 2 mg/m2 Without GCSF | 3 mg/m2 Without GCSF | 4 mg/m2 Without GCSF | 5 mg/m2 Without GCSF | 6 mg/m2 Without GCSF | 7 mg/m2 Without GCSF | 6 mg/m2 With GCSF | 7 mg/m2 With GCSF | 8 mg/m2 With GCSF | 9 mg/m2 With GCSF | 10 mg/m2 With GCSF
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/6 | 0/3 | 0/6 | 3/10 | 1/9 | 1/4 | 1/3 | 0/3 | 1/7 | 3/7
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6 | 3/3 | 6/6 | 10/10 | 8/9 | 4/4 | 3/3 | 3/3 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2 mg/m2 Without GCSF (N=5) | 3 mg/m2 Without GCSF (N=6) | 4 mg/m2 Without GCSF (N=3) | 5 mg/m2 Without GCSF (N=6) | 6 mg/m2 Without GCSF (N=10) | 7 mg/m2 Without GCSF (N=9) | 6 mg/m2 With GCSF (N=4) | 7 mg/m2 With GCSF (N=3) | 8 mg/m2 With GCSF (N=3) | 9 mg/m2 With GCSF (N=7) | 10 mg/m2 With GCSF (N=7)
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphyloccal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heparin-induced thrombocytopenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant plural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg/m2 Without GCSF (N=5) | 3 mg/m2 Without GCSF (N=6) | 4 mg/m2 Without GCSF (N=3) | 5 mg/m2 Without GCSF (N=6) | 6 mg/m2 Without GCSF (N=10) | 7 mg/m2 Without GCSF (N=9) | 6 mg/m2 With GCSF (N=4) | 7 mg/m2 With GCSF (N=3) | 8 mg/m2 With GCSF (N=3) | 9 mg/m2 With GCSF (N=7) | 10 mg/m2 With GCSF (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 4 | 2 | 2 | 1 | 0 | 1 | 5
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 2 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 | 1 | 5 | 5 | 7 | 3 | 1 | 3 | 4 | 5
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 1 | 2 | 2 | 1 | 2 | 3 | 5
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 (0) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 (0) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Visual disturbance (Eye disorders) | 0 (0) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 (0) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 2 | 2
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Asthenia (General disorders) | 0 (0) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Chest discomfort (General disorders) | 0 (0) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 3 | 2 | 2 | 1 | 1 | 4 | 1 | 3 | 1 | 3 | 5
Gait disturbance (General disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 (0) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 (0) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Pain (General disorders) | 0 (0) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 (0) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral coldness (General disorders) | 0 (0) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 1 | 0 | 2 | 3 | 1 | 0 | 1 | 5 | 0
Suprapubic pain (General disorders) | 0 (0) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 (0) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine colour abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 3
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vein discolouration (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor intends to publish the results of the trial in collaboration with the Investigators.